CLINICAL TRIAL: NCT05079802
Title: Clinical and Radiographic Evaluation of Lesion Sterilization and Tissue Repair in Non-vital Primary Molars Using Double Antibiotic Paste With Two Different Vehicles (Randomized Clinical Trial and In Vitro Study)
Brief Title: Clinical & Radiographic Evaluation of LSTR in Non-vital Primary Molars Using Two Different Vehicles
Acronym: LSTR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Abdel Halim, assisting teacher, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED21-7D
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Resorption of Tooth or Root
MeSH Terms: interventions — Propylene Glycol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): study group
  Interventions: Drug: Double antibiotic paste mixed with chitosan nanoparticles
- Group 2 (Other): control group
  Interventions: Drug: Double antibiotic paste mixed with propylene glycol

INTERVENTIONS:
Drug: Double antibiotic paste mixed with chitosan nanoparticles — Lesion sterilization and tissue repair in non-vital primary molars with double antibiotic paste mixed with chitosan nanoparticles gel
  Other Names: DAP mixed with CHNPs
  Arms: Group 1
Drug: Double antibiotic paste mixed with propylene glycol — Lesion sterilization and tissue repair in non-vital primary molars with double antibiotic paste mixed with propylene glycol
  Other Names: DAP mixed with PG
  Arms: Group 2

SUMMARY:
LSTR will be done for primary teeth with significant root resorption needing non-vital pulp therapy to save such teeth for up to 12 months. The first part will be in vitro study to compare the antimicrobial effect of double antibiotic paste mixed with chitosan nanoparticle vs double antibiotic paste mixed with propylene glycol. The second part will be randomized clinical trial comparing the clinical and radiographic success of LSTR in study group where double antibiotic mix is mixed with chitosan nanoparticles and control group where double antibiotic paste is mixed with propylene glycol .

DETAILED DESCRIPTION:
Clinical and Radiographic Evaluation of Lesion Sterilization and Tissue Repair in Non-vital Primary Molars Using Double Antibiotic Paste with Two Different Vehicles (Randomized Clinical Trial and In Vitro Study)

Introduction:

Healthy primary teeth are important for speech, mastication and to maintain the space for their permanent successors developing in the jaw underneath. Teeth with infected root canals, particularly those in which the infection has reached the peri-radicular tissues, are a common problem in the primary dentition. A relatively new biologic approach, lesion sterilization and tissue repair therapy (LSTR) was introduced. It was modified from 3 mix 1:1:1 metronidazole, ciprofloxacin and minocycline to double mix where 1:1 metronidazole and ciprofloxacin are mixed with propylene glycol. It is indicated for primary teeth with significant root resorption (external resorption greater than 1 mm and/ or internal resorption) needing non-vital pulp therapy. It is also indicated when the clinician decides not to extract the tooth with significant preoperative root resorption, LSTR should be the choice over pulpectomy to save such teeth for up to 12 months. Chitosan it is a natural nontoxic, biocompatible, biodegradable polysaccharide with broad antibacterial spectrum (covering gram-negative and gram-positive bacteria as well as fungi), and it has antioxidant and antitumor properties, also it has the ability to form ﬁlm and gel. Chitosan and chitosan nanoparticle can be used as a vehicle for incorporating natural or chemical antimicrobial agents, however, chitosan nanoparticles exhibit a higher antimicrobial activity than chitosan. Also, chitosan nanoparticles have better absorption and penetration into dentinal tubules

Aim of Study:

1. To evaluate the clinical and radiographic outcomes of using double antibiotic paste mixed with chitosan nanoparticles gel vs. double antibiotic paste mixed with propylene glycol in lesion sterilization and tissue repair in non-vital primary molars.
2. Both materials will be compared in terms of ease of handling, time to perform procedure and convenience of application.
3. Comparing the antibacterial effect of double antibiotic paste mixed with chitosan nanoparticles gel vs. that mixed with propylene glycol in vitro.

Methodology:

1. In Vitro Microbiological Study Before the initiation of the clinical trial, an in vitro study will be carried out. A pilot study to assess the antimicrobial effect of double antibiotic paste mixed with a vehicle of chitosan nanoparticles gel of 2 different concentrations (0.3% and 0.5%) in order to determine which is the better concentration to be used in the lesion sterilization and tissue repair.

   A microbiological study will be carried out to compare the antimicrobial effect of double antibiotic paste mixed with the better concentration of chitosan nanoparticles gel according to the pilot study and double antibiotic paste mixed with propylene glycol. Sample size n=14, each group n=7.

   Procedures:

   A swab will be taken from non-vital primary molars with a paper point and it will be inserted in a suitable transporting medium and cultivated in a suitable medium and different bacterial strains will be identified. The strains will then be isolated and cultivated in suitable media. Materials under investigation will be added to identify the inhibition zones diameters.
2. In Vivo Study

A randomized controlled trial, with 1:1 allocation ratio to either study group (group 1) or control group (group 2). Participants will be medically free children, in the age group 4-7 years, having non-vital primary molars with root resorption more than 1 mm that needs to be retained a tooth for up to 12 months that otherwise would be extracted. Sample size: n=36 molars, (group1) n=18 molars where LSTR will be performed with double antibiotic paste mixed with chitosan nanoparticles gel and (group 2) n=18 molars here LSTR will be performed with double antibiotic paste mixed with propylene glycol.

Procedures:

Caries will be removed with a sterile large round high-speed then pulpotomy will be performed and coronal pulp tissue will be removed using a sterile small sharp excavator, followed by irrigation with 1% sodium hypochlorite. Dryness will be done then double antibiotic will be mixed with chitosan nanoparticles gel until a creamy mix is formed then the mix will be placed in the pulp chamber for (group 1), while double antibiotic will be mixed with propylene glycol until a creamy mix is formed, then the mix will be placed in the pulp chamber for the (group 2). The glass ionomer will be injected to fill the pulp chamber and finally the tooth will be restored with a stainless-steel crown. Follow up will be for one year with recall visits at 1, 3, 6 and 12 months.

Clinical outcome: Reduction/absence of pain, no abnormal mobility/ swelling or abscess.

Radiographic outcomes: Decrease or resolution in interradicular radiolucency and decrease/absence of internal resorption.

ELIGIBILITY:
Inclusion Criteria:

1-Non-vital primary molars

1. With root resorption more than 1 mm that needs to be retained a tooth for up to 12 months that otherwise would be extracted
2. Without mobility up to grade I mobility.

Exclusion Criteria:

1. Non-vital primary molars

   1. With perforation into the bifurcation.
   2. Badly broken down.
   3. With no root resorption.
   4. With excessive bone loss in furcation area involving underlying tooth germ.
   5. Nearing exfoliation.
2. Participants that

   1. Have previous history of allergy to the antibiotics used in the study.
   2. Their caregivers do not oblige to signing the informed consent.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes through clinical examination | Follow up will be for one year with recall visits at 1, 3, 6 and 12 months
  No pain. No abnormal mobility. No swelling
Radiographic outcomes by comparing pre and post treatment radiographic pathologic radiolucent area/s size/s | Follow up will be for one year with recall visits at 1, 3, 6 and 12 months
  Decrease in size / absence of interradicular radiolucency. Decrease in size /absence of internal resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Olaa Abdel Geleel, PhD, Study Chair — Ain Shams University

IPD SHARING:
Plan to Share IPD: No